CLINICAL TRIAL: NCT04249154
Title: Postoperative Hypofractionated Radiation Therapy and Hormonal Therapy in Patients With Prostate Cancer: A Phase II Trial
Brief Title: Postop Hypofractionated Radiation Therapy and LHRH in Patients With Prostate Cancer
Acronym: PROMPT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Tolmar Inc. (Industry)
Responsible Party: Principal Investigator, Fabio Cury, Assitant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-126-MUHC
Record Dates: First submitted 2019-08-15; First posted 2020-01-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Eligard; Post-Operative Hypofractionation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — luprolide acetate gel depot; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-op IMRT & hormonal therapy (Other): The protocol is designed to recruit patients who have undergone prostatectomy and high risk features of the disease were found post-operatively or for patients that, after prostatectomy, a PSA rise has been documented will be enrolled in the Phase II trial. Patients will receive Eligard injection 8-12 weeks before starting radiation. The second injection is given 12 weeks after the first one concomitant with radiation therapy.
  Interventions: Drug: Eligard

INTERVENTIONS:
Drug: Eligard — Eligard dose of 22.5mg given, 50Gy in 20 treatments of radiation therapy to start 12 weeks after first injection concurrent with second injection of Eligard
  Other Names: Radiation

SUMMARY:
Prostate cancer is the second most common cancer among Canadian men of which approximately 20-30% present with high-risk tumour characteristic.

Although surgery can be curative in patients evidencing pathological high-risk disease (extracapsular extension, seminal vesicle involvement, positive surgical margins), a large proportion will develop biochemical failure within years from the surgical procedure. The failure rate is even more pronounced in those patients that present with high prostate specific antigen (PSA) levels, pT3 disease, positive margins and Gleason score ≥8 with an estimated 75% failure rate at 10 years.

Post-operative radiotherapy (RT) has been shown in three randomized trials to significantly decrease the biochemical failure rate and in one of the trials a survival benefit was also seen with the addition of post-operative RT and is considered by many investigators standard therapy in patients with pathological high-risks factors even in absence of biochemical failure.

DETAILED DESCRIPTION:
Although RT is known to potentially eradicate microscopic disease localized in the prostatic bed, the current dilemma is whether to deliver RT in the adjuvant setting (defined as the use of RT post-prostatectomy to patients at a higher risk of recurrence because of adverse pathological features prior to evidence of disease recurrence (i.e., with an undetectable PSA) or to use it as an early salvage therapy (defined as the use of RT in patients with rising PSA but no evidence of metastatic disease).

There are several institutional retrospective reports on the use of RT as salvage therapy but no randomized trial has ever been completed. The best evidence available, however, supports early salvage RT as the best strategy to be used to maximize results.

Our own group has shown excellent results using this approach in patients with low and intermediate risk disease and is currently exploring this approach in patients with high-risk disease. Hypofractionated RT offers a more convenient shorter course of treatment, reduces health-costs and appears to be as effective and safe as conventionally fractionated regimens.

This Phase 2 trial will study the potential role of hypofractionated in the post-operative setting in patients with high-risk features with the primary objective of assessing toxicity from this approach.

The use of androgen deprivation therapy in combination with RT in the primary treatment for patients with intermediate or high-risk prostate cancer is well established. The use of androgen suppression in the post-operative setting has been less explored and its definitive role has not been fully explored.

This is a phase II clinical trial to assess the feasibility and overall toxicity of adding one injection of neo-adjuvant hormonal therapy starting 12 weeks before plus Hypofractionated Radiotherapy for four weeks concurrently with another injection of luteinizing hormone-releasing hormone (LHRH) analog in patients with post-operative setting in patients with high-risk features.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven high risk (any of the following risk factors: surgical positive margins; extra-capsular extension; seminal vesicle involvement, Gleason score >7) adenocarcinoma of the prostate after a radical prostatectomy as primary treatment (adjuvant group), with pathologically negative lymph nodes dissection or clinically negative lymph nodes by imaging [pelvic and abdominal computed tomography (CT) scan, or magnetic resonance imaging (MRI)]. Lymphadenectomy is not mandatory. Any type of prostatectomy will be permitted. For this group of patients, the PSA level at time of entry must be below 0.4 ng/ml
* Histologically proven adenocarcinoma after a radical prostatectomy with pathologically negative lymph nodes (lymphadenectomy is not mandatory) or clinically negative lymph nodes by imaging (pelvic and abdominal CT scan, or MRI or) and evidence of biochemical failure (defined as two consecutives rises of the PSA, at any PSA level). PSA upper limit post-prostatectomy must be below 2.0 ng/ml (salvage group). Any type of prostatectomy will be permitted
* Negative bone metastases proven by bone scan. The use of proton emission tomography (PET) fluoride is allowed
* History and physical examination (including digital rectal exam) within 90 days prior of registration
* Adequate marrow reserve defined as: Hemoglobin ≥ 10 g/dl (patients may be transfused in order to achieve this level); Platelets ≥ 100 000 cells/mm3 and a white blood cell count of ≥ 4000 cells/ml3
* AST or ALT <2 x the upper limit of normal
* PSA and testosterone levels within one month of registration Age ≥ 18
* Zubrod Performance Status 0-1
* Patients must sign a study-specific consent form

Exclusion Criteria:

* Previous exposure to androgen deprivation
* Chemotherapy before or after prostatectomy
* Prior pelvic radiotherapy
* Previous malignancies (except non-melanomatous skin cancer) unless disease-free >5 years
* Severe, active medical condition that makes the use of any of the therapies of the study not recommended

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Trial is for prostate cancer.
Enrollment: 77 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Acute Patient Reported Morbidity in genito-urinary and gastrointestinal toxicity | Up to 90 days after the end of radiation treatment
  Number of Participants With Treatment-Related Adverse Events as Assessed by the Common Terminology Criteria for Adverse Events v.5.0 (CTCAE v5.0), Change From Baseline in genito-urinary and gastrointestinal toxicity up to 12 Weeks. Assessments will be collected at baseline and at the end of radiotherapy treatment and in follow-up.

SECONDARY OUTCOMES:
Acute Physician-Reported Morbidity in genito-urinary and gastrointestinal toxicity | Up to 90 days after the end of radiation treatment
  Number of Participants With Treatment-Related Adverse Events as Assessed by the CTCAE v5.0, Change From Baseline in genito-urinary and gastrointestinal toxicity up to 12 Weeks. Assessments will be collected before and at the end of radiotherapy treatment and in follow-up. For each symptom i.e., frequency, severity, the worst score experienced by the patient will be recorded.
Late Patient-Reported Morbidity in genito-urinary and gastrointestinal toxicity | from the end of radiotherapy up to five years
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0, Change From Baseline in genito-urinary and gastrointestinal toxicity. Assessments will be collected at baseline and up to 5 years of follow-up. For each symptom i.e., frequency, severity, the worst score experienced by the patient will be recorded will be collected before and at the end of radiotherapy treatment and in follow-up.

OTHER OUTCOMES:
Late Physician-Reported Morbidity in genito-urinary and gastrointestinal toxicity | From the end of radiation therapy + 90 days to the time of the first recorded late grade 3+ adverse event, assessed up to 5 years
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0, Change From Baseline in genito-urinary and gastrointestinal toxicity. Assessments will be collected at baseline and at the end of 5 years of follow-up. For each symptom i.e., frequency, severity, the worst score experienced by the patient will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Cury, MD, Principal Investigator — Radiation Oncologist
Locations (2):
- Canada (2):
  - McGill University Health Centre- Cedars Cancer Centre, Montreal, Quebec
  - McGill University Health Centre-Cedars Cancer Centre, Montreal, Quebec

REFERENCES:
- [Background] Punnen S, Cooperberg MR. The epidemiology of high-risk prostate cancer. Curr Opin Urol. 2013 Jul;23(4):331-6. doi: 10.1097/MOU.0b013e328361d48e. PMID 23619582
- [Background] Nguyen CT, Reuther AM, Stephenson AJ, Klein EA, Jones JS. The specific definition of high risk prostate cancer has minimal impact on biochemical relapse-free survival. J Urol. 2009 Jan;181(1):75-80. doi: 10.1016/j.juro.2008.09.027. Epub 2008 Nov 13. PMID 19012927
- [Background] Wiegel T, Bartkowiak D, Bottke D, Bronner C, Steiner U, Siegmann A, Golz R, Storkel S, Willich N, Semjonow A, Stockle M, Rube C, Rebmann U, Kalble T, Feldmann HJ, Wirth M, Hofmann R, Engenhart-Cabillic R, Hinke A, Hinkelbein W, Miller K. Adjuvant radiotherapy versus wait-and-see after radical prostatectomy: 10-year follow-up of the ARO 96-02/AUO AP 09/95 trial. Eur Urol. 2014 Aug;66(2):243-50. doi: 10.1016/j.eururo.2014.03.011. Epub 2014 Mar 21. PMID 24680359
- [Background] Thompson IM Jr, Tangen CM, Paradelo J, Lucia MS, Miller G, Troyer D, Messing E, Forman J, Chin J, Swanson G, Canby-Hagino E, Crawford ED. Adjuvant radiotherapy for pathologically advanced prostate cancer: a randomized clinical trial. JAMA. 2006 Nov 15;296(19):2329-35. doi: 10.1001/jama.296.19.2329. PMID 17105795
- [Background] Bolla M, van Poppel H, Tombal B, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Colombel M, van de Beek C, Verhagen P, van den Bergh A, Sternberg C, Gasser T, van Tienhoven G, Scalliet P, Haustermans K, Collette L; European Organisation for Research and Treatment of Cancer, Radiation Oncology and Genito-Urinary Groups. Postoperative radiotherapy after radical prostatectomy for high-risk prostate cancer: long-term results of a randomised controlled trial (EORTC trial 22911). Lancet. 2012 Dec 8;380(9858):2018-27. doi: 10.1016/S0140-6736(12)61253-7. Epub 2012 Oct 19. PMID 23084481
- [Background] Freedland SJ, Rumble RB, Finelli A, Chen RC, Slovin S, Stein MN, Mendelson DS, Wackett C, Sandler HM; American Society of Clinical Oncology. Adjuvant and salvage radiotherapy after prostatectomy: American Society of Clinical Oncology clinical practice guideline endorsement. J Clin Oncol. 2014 Dec 1;32(34):3892-8. doi: 10.1200/JCO.2014.58.8525. Epub 2014 Nov 3. PMID 25366677
- [Background] King CR. Adjuvant versus salvage radiotherapy for high-risk prostate cancer patients. Semin Radiat Oncol. 2013 Jul;23(3):215-21. doi: 10.1016/j.semradonc.2013.01.009. PMID 23763888
- [Background] Spiotto MT, Hancock SL, King CR. Radiotherapy after prostatectomy: improved biochemical relapse-free survival with whole pelvic compared with prostate bed only for high-risk patients. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):54-61. doi: 10.1016/j.ijrobp.2007.02.035. Epub 2007 Apr 24. PMID 17459606
- [Background] Patel N, Faria S, Cury F, David M, Duclos M, Shenouda G, Ruo R, Souhami L. Hypofractionated radiation therapy (66 Gy in 22 fractions at 3 Gy per fraction) for favorable-risk prostate cancer: long-term outcomes. Int J Radiat Oncol Biol Phys. 2013 Jul 1;86(3):534-9. doi: 10.1016/j.ijrobp.2013.02.010. Epub 2013 Apr 15. PMID 23597418
- [Background] Kruser TJ, Jarrard DF, Graf AK, Hedican SP, Paolone DR, Wegenke JD, Liu G, Geye HM, Ritter MA. Early hypofractionated salvage radiotherapy for postprostatectomy biochemical recurrence. Cancer. 2011 Jun 15;117(12):2629-36. doi: 10.1002/cncr.25824. Epub 2010 Dec 14. PMID 21656740
- [Background] Pilepich MV, Winter K, Lawton CA, Krisch RE, Wolkov HB, Movsas B, Hug EB, Asbell SO, Grignon D. Androgen suppression adjuvant to definitive radiotherapy in prostate carcinoma--long-term results of phase III RTOG 85-31. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1285-90. doi: 10.1016/j.ijrobp.2004.08.047. PMID 15817329
- [Background] Hanks GE, Pajak TF, Porter A, Grignon D, Brereton H, Venkatesan V, Horwitz EM, Lawton C, Rosenthal SA, Sandler HM, Shipley WU; Radiation Therapy Oncology Group. Phase III trial of long-term adjuvant androgen deprivation after neoadjuvant hormonal cytoreduction and radiotherapy in locally advanced carcinoma of the prostate: the Radiation Therapy Oncology Group Protocol 92-02. J Clin Oncol. 2003 Nov 1;21(21):3972-8. doi: 10.1200/JCO.2003.11.023. PMID 14581419
- [Background] Bolla M, Van Tienhoven G, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Billiet I, Torecilla JL, Pfeffer R, Cutajar CL, Van der Kwast T, Collette L. External irradiation with or without long-term androgen suppression for prostate cancer with high metastatic risk: 10-year results of an EORTC randomised study. Lancet Oncol. 2010 Nov;11(11):1066-73. doi: 10.1016/S1470-2045(10)70223-0. Epub 2010 Oct 7. PMID 20933466
- [Background] Widmark A, Klepp O, Solberg A, Damber JE, Angelsen A, Fransson P, Lund JA, Tasdemir I, Hoyer M, Wiklund F, Fossa SD; Scandinavian Prostate Cancer Group Study 7; Swedish Association for Urological Oncology 3. Endocrine treatment, with or without radiotherapy, in locally advanced prostate cancer (SPCG-7/SFUO-3): an open randomised phase III trial. Lancet. 2009 Jan 24;373(9660):301-8. doi: 10.1016/S0140-6736(08)61815-2. Epub 2008 Dec 16. PMID 19091394
- [Background] Denham JW, Steigler A, Lamb DS, Joseph D, Mameghan H, Turner S, Matthews J, Franklin I, Atkinson C, North J, Poulsen M, Christie D, Spry NA, Tai KH, Wynne C, Duchesne G, Kovacev O, D'Este C; Trans-Tasman Radiation Oncology Group. Short-term androgen deprivation and radiotherapy for locally advanced prostate cancer: results from the Trans-Tasman Radiation Oncology Group 96.01 randomised controlled trial. Lancet Oncol. 2005 Nov;6(11):841-50. doi: 10.1016/S1470-2045(05)70348-X. PMID 16257791
- [Background] Warde P, Mason M, Ding K, Kirkbride P, Brundage M, Cowan R, Gospodarowicz M, Sanders K, Kostashuk E, Swanson G, Barber J, Hiltz A, Parmar MK, Sathya J, Anderson J, Hayter C, Hetherington J, Sydes MR, Parulekar W; NCIC CTG PR.3/MRC UK PR07 investigators. Combined androgen deprivation therapy and radiation therapy for locally advanced prostate cancer: a randomised, phase 3 trial. Lancet. 2011 Dec 17;378(9809):2104-11. doi: 10.1016/S0140-6736(11)61095-7. Epub 2011 Nov 2. PMID 22056152
- [Background] D'Amico AV, Manola J, Loffredo M, Renshaw AA, DellaCroce A, Kantoff PW. 6-month androgen suppression plus radiation therapy vs radiation therapy alone for patients with clinically localized prostate cancer: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):821-7. doi: 10.1001/jama.292.7.821. PMID 15315996
- [Background] Shipley WU, Hunt D, Lukka H, Major P, Heney NM, Grignon D, et al. Initial Report of RTOG 9601: A Phase III Trial in Prostate Cancer: Anti-androgen Therapy (AAT) with Bicalutamide during and after Radiation Therapy (RT) Improves Freedom from Progression and Reduces the Incidence of Metastatic Disease in Patients following Radical Prostatectomy (RP) with pT2-3, N0 Disease, and Elevated PSA Levels. International Journal of Radiation Oncology • Biology • Physics.78(3):S27.
- [Background] Green HJ, Pakenham KI, Headley BC, Yaxley J, Nicol DL, Mactaggart PN, Swanson C, Watson RB, Gardiner RA. Altered cognitive function in men treated for prostate cancer with luteinizing hormone-releasing hormone analogues and cyproterone acetate: a randomized controlled trial. BJU Int. 2002 Sep;90(4):427-32. doi: 10.1046/j.1464-410x.2002.02917.x. PMID 12175403